CLINICAL TRIAL: NCT07258303
Title: Evaluating Safety and Efficacy of Oral-Spray Bacillus Spore Probiotics (LiveSpo Smile CARE) in Preventing and Supporting the Treatment of Periodontal Diseases in Elderly in Hanoi
Brief Title: Oral-Spray Bacillus Spore Probiotics for Periodontal Disease Prevention and Supprotive Treatment in the Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anabio R&D (Industry)
Collaborators: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TNLS.2025.NC
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Periodontal Disease; Oral Deseases
Keywords: Periodontal Disease; The elderly; pathogenic bacterial densities; Bacillus; Spores; oral-spray probiotics
MeSH Terms: conditions — Periodontal Diseases | interventions — Oral Sprays

STUDY DESIGN:
Intervention Model Description: Blind, randomized, and controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo Smile CARE and placebo are indistinguishable regarding taste and smell. The color and turbidity of LiveSpo Smile CARE suspension are unrecognizable to investigators, trainers, caregivers, and paticipants due to opaque plastic container. Only the independent statistician is aware of the group codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants allocated to the placebo group will receive a 0.9% NaCl physiological saline spray. The solution will be self-administered via spray, twice daily-once in the afternoon and once at night. At each administration, participants will apply two sprays to each side of the dental arch and two sprays to the incisor region, resulting in a total of six sprays per application. This regimen will be maintained consistently for a period of 4 weeks.
  Interventions: Drug: oral-spray 0.9% NaCl physiological saline solution
- Smile Care (Experimental): Participants assigned to the experimental group will receive LiveSpo® Smile CARE (20 mL), formulated as an oral-spray probiotics containing ≥ 1 × 10⁹ CFU/ mL of Bacillus subtilis and Bacillus clausii, of 0.9% sodium chloride solution. The suspension will be self-administered via oral spray twice daily once in the afternoon and once at night. At each administration, participants will apply two sprays to each side of the dental arch and two sprays to the incisor region, totaling six sprays per application. The intervention will be continued for a duration of 4 weeks.
  Interventions: Combination Product: LiveSpo Smile CARE

INTERVENTIONS:
Drug: oral-spray 0.9% NaCl physiological saline solution — The oral-spray 0.9% NaCl physiological saline solution is prepared by extracting 20 mL from a 500 mL polypropylene bottle of 0.9% NaCl intravenous infusion (B. Braun, Germany; product declaration No. VD-32732-19). The solution is contained in an opaque plastic spray bottle identical to that used for the administration of Smile Care.
  Other Names: Registration number: VD-32723-19
  Arms: Placebo
Combination Product: LiveSpo Smile CARE — LiveSpo Smile CARE is manufactured as a Class-A medical device (product declaration 250002196/PCBA-HN) in compliance with manufacturing standards approved by the Hanoi Department of Health, Ministry of Health. The product is formulated as a 0.9% NaCl physiological saline solution plus Bacillus subtilis ANA48 and Bacillus clausii ANA39 at total concentration of ≥ 1 billion CFU/ (20 billion CFU/20 mL suspension)
  Arms: Smile Care

SUMMARY:
Periodontal diseases are strongly associated with dysbiosis of the oral microbiome within the biofilm. Key pathogens, including Streptococcus mutans, Aggregatibacter actinomycetemcomitans, and Porphyromonas gingivalis, contribute to caries progression and periodontal inflammation. Given the limitations of antibiotic use and their potential side effects, probiotics represent a promising biological approach to restore microbial balance and support oral health.

In this study, researchers propose that direct application of probiotic spray into the oral cavity is safe and effective in alleviating typical symptoms of periodontal disease, particularly by reducing pathogenic bacterial density.

The objective of this study is to evaluate the safety and efficacy of a oral-spray Bacillus spore probiotics (LiveSpo Smile CARE), containing Bacillus subtilis ANA48 and Bacillus clausii ANA39 at a concentration of ≥ 1 billion CFU/mL x 20 mL formulation, for the prevention and supportive treatment of periodontal disease.

Study Design:

* Sample Size: 90 participants
* Study Location: an elderly care center in Hanoi, Vietnam

Intervention Description: A total of 90 eligible participants will be randomly assigned to two groups (n = 45 per group).

* The Placebo Group will receive 0.9% NaCl physiological saline, spray twice daily (afternoon and evening), with two sprays per application at three sites (both dental arches and the front teeth), totaling six sprays per use, for four consecutive weeks.
* The Smile Care Group will receive an oral-spray probiotics containing ≥ 1 billion CFU/mL × 20 mL of Bacillus subtilis and Bacillus clausii (LiveSpo Smile CARE), administered with the same dosage and frequency as the placebo group.

All participants will receive blinded, coded spray bottles to ensure objectivity. Both groups will be instructed to use the same standardized toothpaste during the study period. Caregivers will monitor the health status of participants and record relevant information in their medical records. During the study, caregivers will be instructed not to provide any additional probiotic oral care products or the solution contains similar components.

Study Duration: 12-18 months.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), severe oral disease is estimated to affect over 1 billion individuals worldwide. Studies have demonstrated that the prevalence of periodontal disease increases with age. In Vietnam, oral disease is a common oral health problem among the elderly, with a prevalence rate of approximately 91%. This includes 51.6% presenting with simple gingivitis and 39.4% with periodontitis. If left untreated, oral disease may lead to gingival inflammation, swelling, bleeding, and destruction of the supporting structures of the teeth, resulting in pain during mastication. In severe cases, it can cause tooth loss, systemic infections such as sepsis, and increase the long-term risk of systemic diseases including cardiovascular disease and diabetes.

Conventional treatment primarily focuses on the mechanical removal of dental plaque through tooth brushing and flossing. While these methods are effective in reducing gingival inflammation and bacterial load, they often fail to completely eliminate plaque, especially in interdental areas. Probiotics have shown promising potential as adjunctive therapy in the management of periodontal disease by restoring microbial balance, modulating host inflammatory responses, and reducing the levels of pathogenic bacteria.

The objective of this study is to evaluate the prevention and supportive therapeutic efficacy of a oral-spray Bacillus spore probiotics (LiveSpo Smile CARE) in alleviating typical symptoms of periodontal disease. Investigators will assess safety, clinical symptom improvement, and reduction in the oral pathogenic bacterial load in elderly participants after 7, 14, 28, and 42 days of using LiveSpo Smile CARE.

This will be a randomized, blind, placebo-controlled clinical trial. The trial will have 12-18 months of duration. Participants will be required to provide demographic data, oral health history, and information regarding prior antibiotic use. Upon providing written informed consent and meeting eligibility criteria, 90 participants will be enrolled and randomly assigned to two groups (n = 45 per group). The placebo group will receive a 0.9% NaCl physiological saline spray, while the intervention group ("Smile Care") will receive the oral-spray probiotics, LiveSpo Smile CARE.

-Primary outcomes

Changes in clinical symptoms (For example: Debris Index-Simplified [DI-S], Gingival Index [GI], Bleeding on Probing [BOP], Gingival Recession [REC], Probing Depth [PD], Clinical Attachment Level [CAL], Halitosis...) at day 28 vs. day 0.

-Secondary outcomes

Changes in cytokine levels (ELISA) and semi-quantification of bacterial pathogens (real-time PCR) in gingival crevicular fluid samples, collected at day 28 compared with day 0.

- Expected outcomes Change in the oral microbiome composition at day 28 vs. day 0.

Presence of Bacillus subtilis ANA48 and Bacillus clausii ANA39 in gingival fluid will be assessed by real-time PCR at follow-up visits (days 7, 14, 28 and 42) compared with day 0, to confirm product use compliance.

Statistical analysis will be conducted using the chi-square test or Fisher's exact test for categorical variables, and t-test, Mann-Whitney test, or Wilcoxon test for continuous variables, depending on data distribution.

ELIGIBILITY:
Inclusion Criteria

* Patients aged 35 years and older.
* Patients diagnosed with periodontal disease based on clinical examination, including gingivitis and periodontitis.
* Patients presenting with at least 10 natural teeth in the dental arch.
* Patients with stable general health status and able to comply with study procedures.
* Patients (or their legal guardians) who provide written informed consent and voluntarily agree to participate in the study.

Exclusion Criteria

* Patients with unstable general health, acute systemic or oral diseases, or malignant conditions that may interfere with participation.
* Patients who are currently receiving treatment for periodontal disease at specialized dental facilities.
* Patients currently using any therapeutic or adjunctive products for the management of periodontal disease.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Oral health indicators | Days 0, 7, 14, 28 and 42
  Percentage of teeth classified according to a grading scale (good, moderate, and severe) for the following parameters: Simple Debris Index (DI-S), Gingival Index (GI), Bleeding on Probing (BOP), and Halitosis (score 1-4) is assessed at various time points relative to day 0.
Periodontal parameters | Days 0, 7, 14, 28 and 42
  Periodontal parameters are assessed for the following: Recession of the Gingival Margin (REC, mm), Probing Depth (PD, mm), and Clinical Attachment Loss (CAL, mm). These parameters are assessed at various time points relative to day 0.

SECONDARY OUTCOMES:
Changes in pro-inflammatory cytokine and IgA levels in gingival crevicular fluid samples at days 0, 7, 14, 28, and 42 | Days 0, 7, 14, 28, and 42
  Changes in pro-inflammatory cytokine levels (e.g. IL-6, IL-8, TNF-alpha...) in gingival crevicular fluid samples.
Changes in the concentration of pathogenic bacteria around the teeth | Days 0, 7, 14, 28, and 42
  Changes in the levels of pathogenic bacteria (P. gingivalis, A. actinomycetemcomitans, and S. mutans) in swab samples taken around the teeth will be evaluated at various time points relative to day 0.

OTHER OUTCOMES:
Changes in the oral microbiome at day 28 compared to day 0 | Days 0 and 28
  Changes in diversity indices and relative taxonomy compositions (16S rRNA NGS) of gingival crevicular fluid samples at day 28 compared to day 0.

CONTACTS AND LOCATIONS:
Overall Officials: Nga TT Pham, PhD. MD, Study Chair — Hanoi Medical University; Thu TH Nguyen, Assoc. Prof., Principal Investigator — Hanoi Medical University; Anh TV Nguyen, Assoc. Prof., Principal Investigator — Spobio Research Center, Anabio R&D
Locations (1):
- Tuyet Thai Senior Care Center, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), and clinical study reports (CSR). For more information or to submit a request, please contact anabio.rd2021@gmail.com

REFERENCES:
- [Result] Berry-Kravis E, Ciurlionis R. Overexpression of fragile X gene (FMR-1) transcripts increases cAMP production in neural cells. J Neurosci Res. 1998 Jan 1;51(1):41-8. doi: 10.1002/(SICI)1097-4547(19980101)51:13.0.CO;2-L. PMID 9452307
- [Result] Jindal G, Pandey RK, Agarwal J, Singh M. A comparative evaluation of probiotics on salivary mutans streptococci counts in Indian children. Eur Arch Paediatr Dent. 2011 Aug;12(4):211-5. doi: 10.1007/BF03262809. PMID 21806906
- [Result] Dang HT, Tran DM, Phung TTB, Bui ATP, Vu YH, Luong MT, Nguyen HM, Trinh HT, Nguyen TT, Nguyen AH, Van Nguyen AT. Promising clinical and immunological efficacy of Bacillus clausii spore probiotics for supportive treatment of persistent diarrhea in children. Sci Rep. 2024 Mar 18;14(1):6422. doi: 10.1038/s41598-024-56627-9. PMID 38494525
- [Result] Aleti G, Sessitsch A, Brader G. Genome mining: Prediction of lipopeptides and polyketides from Bacillus and related Firmicutes. Comput Struct Biotechnol J. 2015 Mar 24;13:192-203. doi: 10.1016/j.csbj.2015.03.003. eCollection 2015. PMID 25893081
- [Result] Bader J, Albin A, Stahl U. Spore-forming bacteria and their utilisation as probiotics. Benef Microbes. 2012 Mar 1;3(1):67-75. doi: 10.3920/BM2011.0039. PMID 22348911
- [Result] Graves D. Cytokines that promote periodontal tissue destruction. J Periodontol. 2008 Aug;79(8 Suppl):1585-91. doi: 10.1902/jop.2008.080183. PMID 18673014
- [Result] Fontana M, Zero DT. Assessing patients' caries risk. J Am Dent Assoc. 2006 Sep;137(9):1231-9. doi: 10.14219/jada.archive.2006.0380. PMID 16946427
- [Result] Teughels W, Durukan A, Ozcelik O, Pauwels M, Quirynen M, Haytac MC. Clinical and microbiological effects of Lactobacillus reuteri probiotics in the treatment of chronic periodontitis: a randomized placebo-controlled study. J Clin Periodontol. 2013 Nov;40(11):1025-35. doi: 10.1111/jcpe.12155. Epub 2013 Sep 15. PMID 24164569
- [Result] Amaliya A, Laine ML, Delanghe JR, Loos BG, Van Wijk AJ, Van der Velden U. Java project on periodontal diseases: periodontal bone loss in relation to environmental and systemic conditions. J Clin Periodontol. 2015 Apr;42(4):325-32. doi: 10.1111/jcpe.12381. Epub 2015 Mar 24. PMID 25683157
- [Result] Hajishengallis G, Lamont RJ. Beyond the red complex and into more complexity: the polymicrobial synergy and dysbiosis (PSD) model of periodontal disease etiology. Mol Oral Microbiol. 2012 Dec;27(6):409-19. doi: 10.1111/j.2041-1014.2012.00663.x. Epub 2012 Sep 3. PMID 23134607
- [Result] Perez-Chaparro PJ, Duarte PM, Shibli JA, Montenegro S, Lacerda Heluy S, Figueiredo LC, Faveri M, Feres M. The Current Weight of Evidence of the Microbiologic Profile Associated With Peri-Implantitis: A Systematic Review. J Periodontol. 2016 Nov;87(11):1295-1304. doi: 10.1902/jop.2016.160184. Epub 2016 Jul 15. PMID 27420109
- [Result] Perez-Chaparro PJ, Goncalves C, Figueiredo LC, Faveri M, Lobao E, Tamashiro N, Duarte P, Feres M. Newly identified pathogens associated with periodontitis: a systematic review. J Dent Res. 2014 Sep;93(9):846-58. doi: 10.1177/0022034514542468. Epub 2014 Jul 29. PMID 25074492